CLINICAL TRIAL: NCT05604898
Title: A Phase 2，Multicenter, Randomized, Double-blind, Placebo-controlled，Multiple-dose Escalation and Dose Finding Study to Evaluate the Safety，PK and Efficacy of Recombinant Anti-IL-17A Humanized Monoclonal Antibody in Chinese Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Phase 2 Study of Recombinant Anti-IL-17A Humanized Monoclonal Antibody in Chinese Participants With Moderate-to-Severe Plaque Psoriasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ -608- Psoriasis-II-01
Record Dates: First submitted 2022-10-31; First posted 2022-11-03 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part 1：608 40 mg (Experimental): Randomized in a 6:2 ratio to 608 40mg or placebo 2-weekly by subcutaneous injection during induction period. During the maintenance period, participants will receive 608 40mg or placebo 4-weekly.
  Interventions: Drug: Recombinant Anti-IL-17A Humanized Monoclonal Antibody Injection; Other: Placebo
- Part 1：608 80 mg (Experimental): Randomized in a 10:2 ratio to 608 80mg or placebo 2-weekly by subcutaneous injection during induction period. During the maintenance period, participants will receive 608 80mg or placebo 4-weekly.
  Interventions: Drug: Recombinant Anti-IL-17A Humanized Monoclonal Antibody Injection; Other: Placebo
- Part 1：608 160 mg (Experimental): Randomized in a 10:2 ratio to 608 160mg or placebo 2-weekly by subcutaneous injection during induction period. During the maintenance period, participants will receive 608 160mg or placebo 4-weekly.
  Interventions: Drug: Recombinant Anti-IL-17A Humanized Monoclonal Antibody Injection; Other: Placebo
- Part 2：608 160 mg W0+80 mg Q2W+80 mg Q4W (Experimental): Participants will receive starting dose of 160 mg 608 at week 0 followed by 80mg 608 once every two weeks (Q2W) by subcutaneous injection during induction period. During the maintenance period, participants will receive 80mg 608 once every four weeks (Q4W).
  Interventions: Drug: Recombinant Anti-IL-17A Humanized Monoclonal Antibody Injection; Other: Placebo
- Part 2：608 160 mg Q2W+160 mg Q4W (Experimental): Participants will receive 160mg 608 once every two weeks (Q2W) by subcutaneous injection during induction period followed by 160mg 608 once every four weeks (Q4W) during maintenance period.
  Interventions: Drug: Recombinant Anti-IL-17A Humanized Monoclonal Antibody Injection
- Part 2：608 160 mg Q4W+160 mg Q8W (Experimental): Participants will receive 160mg 608 once every four weeks (Q4W) by subcutaneous injection during induction period followed by 160mg 608 once every eight weeks (Q8W) during maintenance period.
  Interventions: Drug: Recombinant Anti-IL-17A Humanized Monoclonal Antibody Injection; Other: Placebo
- Part 2：Placebo (Placebo Comparator): Participants will receive Placebo by subcutaneous injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Recombinant Anti-IL-17A Humanized Monoclonal Antibody Injection — 608 will be administered subcutaneously.
  Other Names: 608
  Arms: Part 1：608 160 mg; Part 1：608 40 mg; Part 1：608 80 mg
Other: Placebo — Participants will receive Placebo to maintain the blinding of the Investigational Medicinal Products.
  Other Names: PBO
  Arms: Part 1：608 160 mg; Part 1：608 40 mg; Part 1：608 80 mg
Drug: Recombinant Anti-IL-17A Humanized Monoclonal Antibody Injection — 608 will be provided at pre-specified time intervals.
  Other Names: 608
  Arms: Part 2：608 160 mg Q2W+160 mg Q4W; Part 2：608 160 mg Q4W+160 mg Q8W; Part 2：608 160 mg W0+80 mg Q2W+80 mg Q4W
Other: Placebo — Participants will receive Placebo at pre-specified time points to maintain the blinding of the Investigational Medicinal Products.
  Other Names: PBO
  Arms: Part 2：608 160 mg Q4W+160 mg Q8W; Part 2：608 160 mg W0+80 mg Q2W+80 mg Q4W; Part 2：Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of the study drug recombinant anti-IL-17A humanized monoclonal antibody in Chinese participants with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
Study SSGJ-608-PsO-II-01 is a phase 2, multicenter, randomized, double-blind, placebo-controlled, multiple-dose escalation and dose finding study to identify the doses of treatments ，and to further evaluate the effect of different dose regimens of recombinant anti-IL-17A humanized monoclonal antibody versus placebo in Chinese participants with moderate-to-severe plaque psoriasis during an induction dosing period with dosing for 12 weeks, followed by a randomized, double-blind, 40-week maintenance dosing period. Phase Ib One of three dose levels of copanlisib is assigned at registration according to the dose escalation scheme. Phase II The copanlisib dose for the Phase II part of the trial will be based on the MTD established in the Phase Ib part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 Years to 65 Years, both male and female.
* BMI ≥18 kg/m^2 and ≤32 kg/m^2 ，and male weight ≥50 kg, female weight ≥45 kg during the screening.
* Chronic plaque psoriasis (PSO) for at least 6 months prior to the randomizationas as determined by the investigator..
* Psoriasis Area Severity Index (PASI) >=12 and body surface area (BSA) affected by PSO >=10% and Static Physician Global Assessment (sPGA) score >=3.
* According to the judgment of the investigator, the subject needs to receive systemic treatment and / or phototherapy (including subjects who have used local treatment, and / or phototherapy, and / or poor control of previous systemic treatment).
* Subject must be able to understand and comply with the requirements of the study. and must participate voluntarily and sign the written informed consent.

Exclusion Criteria:

* History of pustular or erythrodermic psoriasis other than plaque psoriasis at screening or baseline.
* History of drug-induced psoriasis.
* Ongoing use of prohibited treatments.
* Have previously received any drug that directly targets IL-17.
* Have concurrent or recent use of any biologic agent within washout periods or <5 half-lives prior to randomization.
* Chronic infections including HIV, viral hepatitis (hepatitis B, hepatitis C), syphilis and/ or active tuberculosis.
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse event (TEAE). | Up to 64 Weeks
  The incidence and severity of treatment emergent adverse event (TEAE), including adverse events (AEs)，serious adverse event (SAE) and AEs associated with the use of the drug, as well as clinical symptoms, and any abnormalities of vital signs, physical examinations，electrocardiogram，laboratory tests and, etc.

SECONDARY OUTCOMES:
Cmax | Week 0 to 16
  To assess the maximum plasma level of 608.
Tmax | Week 0 to 16
  To assess the time to peak 608 concentration.
AUC0-last | Week 0 to 16
  To assess the area under the concentration time-curves from time zero to the time of the last quantifiable concentration after dosing.
AUC0-tau | Week 0 to 16
  To assess the area under the concentration time-curves from time zero to the dosing interval tau.
Cmin | Week 0 to 48
  To assess the minimum plasma level of 608.
Rac_Cmax | week 0,12
  Accumulation ratio based on maximum plasma concentration (Cmax) calculated as: Rac_Cmax = Cmax at steady state (ss) divided by Cmax at first dose.
Rac_AUC0-tau | week 0,12
  Accumulation ratio calculated as, Rac obtained from Area Under the Concentration Time Curve (AUCτau) from time 0-τau（Week 12） divided by AUC from time 0-τau （Week 0）
Number of Participants Positive for Anti-Drug Antibody (ADA) in Part 1. | Week 0,4,8,12,16,24,48,64
  Serum ADA positivity is determined over course of the trial duration.
Number of Participants Positive for Anti-Drug Antibody (ADA) in Part 2. | Week 0,8,20,44,64
  Serum ADA positivity is determined over course of the trial duration.
Percentage of Participants Achieving a ≥75% Improvement in Psoriasis Area and Severity Index (PASI 75) | At Week 12
  The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs(0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Percentage of Participants With a Static Physician Global Assessment (sPGA) Score of Clear (0) or Minimal (1) With at Least a 2 Point Improvement | At Week 12
  The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participants Ps were assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe). An sPGA responder was defined as having a postbaseline sPGA score of "0" or "1" with at least a 2-point improvement from baseline.
Percentage of Participants Achieving a ≥90% Improvement in Psoriasis Area and Severity Index (PASI 90) | At Week 12
  The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs(0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Percentage of Participants Achieving a 100% Improvement in Psoriasis Area and Severity Index (PASI 100) | At Week 12
  The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs(0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Xu, MD, Principal Investigator — Shanghai Huanshan Hospital Fudan University-Dermatology
Locations (3):
- China (3):
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No